CLINICAL TRIAL: NCT04552444
Title: Clinical Efficacy of Combination Therapy Based on High-dose Biapenem in CRKP Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Man Huang, Ph.D, Sponsor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: SAHZU2017087
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: High-dose Biapenem
Keywords: High-dose Biapenem; Carbapenem resistance Klebsiella pneumoniae; Clinical Efficacy
MeSH Terms: interventions — biapenem

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Klebsiella pneumoniae isolated from sputum, urine and feces of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the death group: Through the corresponding treatment, the patients who died within 28 days
  Interventions: Drug: Biapenem
- the survival group: Through the corresponding treatment, the patients who survived within 28 days
  Interventions: Drug: Biapenem

INTERVENTIONS:
Drug: Biapenem — In the course of CRKP treatment, double dose biapenem was selected.

SUMMARY:
Carbapenem resistance is a high mortality rate of Klebsiella pneumoniae infection. It has been proved that high-dose carbapenem can reduce mortality and has a certain clinical effect. In this study, a high dose of biapenem was compared to determine whether it had a similar effect than meropenem.

ELIGIBILITY:
Inclusion Criteria:

* ICU hospitalized for more than 3 days;
* Biapenem used for more than 3 days

Exclusion Criteria:

* Patients who refuse to be included in the group or pregnant women or under the age of 14 or ICU hospitalized for less than 3 days

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Most of the patients were from the coastal areas of the Yangtze River, and some of them were exposed to all parts of the country.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 2017.01.01-2021.12.31

SECONDARY OUTCOMES:
Clearance rate of pathogenic microorganisms | 2017.01.01-2021.12.31
ICU hospitalization days | 2017.01.01-2021.12.31

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Please Select, China

IPD SHARING:
Plan to Share IPD: Undecided